CLINICAL TRIAL: NCT05263570
Title: The Efficiency for Patient With Stage II-III HR+/HER2+ Early Breast Cancer With Standard Neoadjuvant Therapy: a Retrospective, Multicenter Study in Real World Settings.
Brief Title: The Efficiency for Stage II-III HR+/HER2+ Early Breast Cancer Patient With Standard Neoadjuvant Therapy in Real World.
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Professor, Shengjing Hospital
Other Study IDs: HR-HER2-RWS-01
Record Dates: First submitted 2022-01-17; First posted 2022-03-02 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
Keywords: standard Therapy （TCbHP/THP/EC-THP/AC-THP）
MeSH Terms: conditions — Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage II-III HR+/HER2+ Early Breast Cancer: Stage II-III HR+/HER2+ Early Breast Cancer
  Interventions: Drug: Standard Therapy

INTERVENTIONS:
Drug: Standard Therapy — Standard Therapy, including TCbHP, THP, EC-THP, AC-THP
  Other Names: TCbHP, THP, EC-THP, AC-THP

SUMMARY:
To observe the efficiency for patient with stage II-III HR+/HER2+ early breast cancer with standard neoadjuvant therapy, a retrospective, multicenter study in real world settings.

DETAILED DESCRIPTION:
This study collected patients used standard neoadjuvant therapy (TCbHP/THP/EC-THP/AC-THP) among stage II-III HR+/HER2+ early breast cancer, and to describe patient clinical characteristics and clinical outcomes of them in real world settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or older
* HR+/HER2- breast cancer diagnosis based on local standards
* Women having stage II-III breast cancer diagnosed based on AJCC cancer staging system (8th edition) who will be admitted because of breast cancer for the first time
* Standard Therapy, determined at the discretion of the investigator, including （TCbHP/THP/EC-THP/AC-THP）
* Complete medical history was available
* Karnofsky Performance Status (KPS) Scale score ≥ 70

Exclusion Criteria:

* Women who have received any form of anti-tumor treatment - (chemotherapy, radiotherapy, molecular targeted therapy, or endocrine therapy)
* Pregnant or breast-feeding women
* Those who have bilateral breast cancer, inflammatory breast cancer or occult breast cancer
* Those who have stage IV breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stage II-III HR+/HER2+ early breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR) | through study completion, an average of 1 year
  tpCR is defined as the absence of residual invasive cancer on resected breast specimen and the sampled regional lymph nodes as shown by hematoxylin-eosin staining after completion of the neoadjuvant treatment.

SECONDARY OUTCOMES:
Best overall response rate (BORR) [ Time Frame: During neoadjuvant treatment | through study completion, an average of 1 year
  The proportion of patients who respond to the treatment at any study time point
Residual cancer burden (RCB) | through study completion, an average of 1 year
  RCB score is obtained according to pathological evaluation after completion of neoadjuvant treatment and surgery

OTHER OUTCOMES:
Overall survival (OS) | Within 5 years after surgery
  It refers to the length of time from the start of treatment to the death of the patient.
Disease-free survival (DFS) | Within 5 years after surgery
  It refers to the length of time from the start of medication after enrollment to the death of the patient because of the recurrence, distant metastasis of the disease, invasive contralateral breast cancer, or any other cause.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, PHD, Study Chair — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided